CLINICAL TRIAL: NCT02421614
Title: Effect of Enteral Feeding's Macronutrient Composition on Inflammatory Mediators, Oxidative Stress and Outcomes in Intensive Care Unit Patients With Acute Respiratory Failure
Brief Title: Enteral Feeding Composition and Acute Respiratory Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zahra Vahdat Shariatpanahi (Other)
Responsible Party: Sponsor-Investigator, Zahra Vahdat Shariatpanahi, Assistant professor, Shahid Beheshti University
Organization: Shahid Beheshti University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 054575
Record Dates: First submitted 2015-04-07; First posted 2015-04-20 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-11

CONDITIONS: Acute Respiratory Failure
Keywords: acute respiratory failure; lung; enteral feeding; feeding composition; olive; high fat
MeSH Terms: interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- high olive oli (Experimental): A high fat (45%) low carbohydrate (35%) enteral feeding will be administered to acute respiratory failure patients. The percentage of olive oil will be half of total fat.
  Interventions: Other: high-protein low-carbohydrate diet with high olive oil
- high sunflower oil (Experimental): A high fat (45%) low carbohydrate (35%) enteral feeding will be administered to acute respiratory failure patients. The total fat will be sunflower oil.
  Interventions: Other: high-protein low-carbohydrate diet with high sunflower oil
- kitchen formula (No Intervention): A high protein kitchen diet for tube feeding will be administered to acute respiratory failure patients.

INTERVENTIONS:
Other: high-protein low-carbohydrate diet with high olive oil
  Arms: high olive oli
Other: high-protein low-carbohydrate diet with high sunflower oil
  Arms: high sunflower oil

SUMMARY:
This study aimed to investigate the effect of enteral feeding's macronutrient composition on inflammatory mediators, oxidative stress and outcomes in Intensive Care Unit (ICU) patients with acute respiratory failure. In this double-blind randomized control trial, 42 patients of both sexes and diagnosed with acute respiratory failure in ICU that receive enteral feeding, will be randomly assigned to three groups of 14 each. First Intervention group; high-protein low-carbohydrate diet with high olive oil, the second intervention group; high-protein low-carbohydrate diet with high sunflower oil and control; high-protein kitchen formula. Intravenous levels of uric acid, high sensitive C-Reactive Protein (hs-CRP), Interleukin 6 (IL-6) and Total Antioxidant Capacity (TAC) measured at days 0 and 10. As well as, organ failure, duration of ventilation, length of ICU stay and mortality rates will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in ICU
* age older than 18 years old
* need to be mechanically ventilation
* have enteral feeding
* no previous diabetes
* no previous HIV infection
* no previous nervous system
* no previous liver failure
* no previous nephrotic syndrome
* not passed more than 48 hours from diagnose of acute respiratory failure

Exclusion Criteria:

* death at less than three days of enteral feeding administration
* extubation at less than three days of enteral feeding administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
length of ventilation | The number of days at least 3, to which days that patient extubated
  The number of days from the patient intubation to his/her extubation

SECONDARY OUTCOMES:
Levels of high sensitive C-Reactive Protein (hs-CRP) in patient's vein blood | 10 days
Levels of Total Antioxidant Capacity (TAC) in patient's vein blood | 10 days
Levels of uric acid in patient's vein blood | 10 days
Levels of Interleukin 6 (IL-6) in patient's vein blood | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nutrition Sciences and Food Technology, Tehran, Iran